CLINICAL TRIAL: NCT04461652
Title: The Drainage Effect of a Chest Tube Plus Prophylactic Air-extraction Catheter vs Traditional Drainage Strategy in Uniportal Upper Lung Lobectomy
Brief Title: The Effect of a Combined Drainage Strategy in Uniportal Upper Lung Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, Associate professor, Tongji University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TongiU
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Cancer; video-assisted thoracic surgery; drainage tube
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, non-inferiority trial, two different drainage strategy will be performed, and both were used routinely in clinical practice. One should be one thoracic tube (28fr drainage tube) was inserted through intercostal incision, and one microtubule (7fr × 20cm) was punctured through the middle line of clavicle, and another will be two conventional chest tubes (28fr or 24fr) were placed through intercostal incision.
Who Masked: Outcomes Assessor
Masking Description: Data collected from the X-rays and the pain score evaluation will be masked and the outcomes assessor have no method to get randomized information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New method (Experimental): One thoracic tube (28fr drainage tube) was inserted through intercostal incision, and one microtubule (7fr × 20cm) was punctured through the middle line of clavicle
  Interventions: Procedure: prophylactic air-extraction catheter drainage
- Traditional method (Placebo Comparator): Two conventional chest tubes (28fr or 24fr) were placed through intercostal incision
  Interventions: Procedure: prophylactic air-extraction catheter drainage

INTERVENTIONS:
Procedure: prophylactic air-extraction catheter drainage — This is a kind of venous catheter commonly used in clinic. It may bring less pain after being inserted into the chest, with an equivalent drainage effect with traditional thick drainage tube from our experience, especially in the aspect of gas drainage effect.

SUMMARY:
Traditional drainage for uniportal video assisted thoracoscopic surgery (VATS) is a routine method, usually with one or two chest tubes at intercostal incisions, but postoperative pain due to the chest tube and unsatisfied drainage effect was noted.

In this study, the investigators are going to explore whether a prophylactic air-extraction catheter combined with chest tube drainage may not increase complications in uniportal VATS for upper lung lobectomy. The patients would be assigned to two arms, one with a prophylactic air-extraction catheter combined with chest tube, and another with two chest tubes, and the effect of the combined drainage strategy will be evaluated.

DETAILED DESCRIPTION:
Research purpose and background:

Surgical resection is still one of the most important treatment methods for early stage non-small cell lung cancer. Complete resection and reasonable dissection of mediastinal lymph nodes are the key of cancer cure. Lobectomy has always been the standard surgical method for lung cancer radical resection. It can remove the lesion and retain normal lung function by resecting the lung lobe where the lesion is and preserve the remaining lobe. In recent years, the development of uniport video-assisted thoracic surgery (VATS) has further reduced the trauma, with treatment benefit similar with that of two-port and three-port thoracoscopy. However, based on the single hole thoracoscopic lung recruitment, incision drainage and other issues also need further evidence support.

No tube technology, such as no tracheal intubation, drainage tube, nor catheter combined with video-assisted thoracoscopy, can significantly improve the rehabilitation of patients, and further shorten the postoperative hospital stay. In addition, the safety of tubeless drainage has been supported by more and more studies. However, poor drainage may also increase the incidence of pneumothorax and postoperative pulmonary dysfunction.

After upper lobe lobectomy, the cavity needs to be filled by the full recruitment of the remaining lobes. theoretically, there is a higher demand for the strategy of the drainage tube. The investigatorstried to compare the safety and effectiveness of the prophylactic air-extraction catheter (later known as microtubule) combined with thoracic tube drainage with traditional double drainage tube alone. Therefore, the investigators conducted a prospective, randomized, non inferiority trial to verify the hypothesis that microtubule combined with thoracic catheter drainage after uniport VATS upper lobectomy will not increase the related perioperative complications compared with traditional thoracic tube drainage.

Quality assurance plan:

1. The doctors participating in the operation and catheterization in clinical trials should be at least attendings, so as to ensure the safety of operation and chest tube placement.
2. The chest tube placement was carried out randomly with two arms.
3. From our previous clinical experience, the tube is placed for 3 days to 2 weeks, so it last for a short time, and all of them can be extubated by doctors above the attending level, so the detachment rate of the experiment is low and the quality can be guaranteed.
4. The trial team has written the test related procedures into the team medical process, including but not limited to the time point of chest X-ray.

Data checks:

Data checks will be performed by a individual attending doctor with GCP to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification:

Source data verification will be performed by a individual attending doctor with GCP to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (for example, medical records, paper or electronic case report forms, or interactive voice response systems).

Data dictionary:

video assisted thoracoscopic surgery, VATS prophylactic air-extraction catheter, PAEC Randomized clinical trial, RCT Non small cell lung cancer, NSCLC

Standard Operating Procedures:

Patients recruitment The subjects were recruited on a voluntary basis. If they decide to participate in this study, the personal data of subjects participating in the trial are confidential. The subject's blood samples will be identified by the study number, not the subject's name. Information that identifies the subject will not be disclosed to members outside the study team unless permission is obtained from the subject. All study members and study sponsors were asked to keep their identities confidential. The subjects' files will be kept in a locked file cabinet for researchers' reference only. In order to ensure that the study is carried out in accordance with the regulations, members of the government administration or the ethics review committee may access the subject's personal data in the research unit as required. At the time of publication, no personal information will be disclosed.

data collection All the patients learned about the two kinds of operation through preoperative education, and voluntarily joined the research group and signed the ethical agreement. In this clinical trial, patients were enrolled in the randomized controlled trial. The members of the experimental group were only responsible for the inclusion and exclusion of patients. The surgeons and assistants did not participate in the preoperative evaluation and postoperative management. The pain assessment team, postoperative management personnel and follow-up evaluators did not know what group the patients belonged to (patients could wear wide clothes to cover the drainage tube after operation)

change management In cases with serious medical risk caused by the operation technology of the trial, or the research indicates that the difference between the groups is too obvious, the researcher should stop the trial and fill in the report form of violation of protocol deviation and report to the ethics committee.

If the patients were enrolled normally and reached the number of cases required for the trial, the trial was finished.

reporting for adverse events

1. The sponsor shall provide the safety research data of the technology and other safety related information.
2. In the design scheme, the definition of adverse events should be clearly defined, and the criteria for judging the severity of adverse events, as well as the classification criteria for judging the relationship between adverse events and experimental operation (such as positively related, possibly related, possibly unrelated, irrelevant and unable to be determined). The protocol requires researchers to truthfully fill in the adverse event record form, recording the occurrence time, severity, duration, measures taken and outcome.
3. Before starting the trial, the members of the research team must be familiar with the contents of the prevention and treatment of subjects and emergency plans in medical treatment.
4. In case of SAE, the research physician must report to the project leader, the food and drug administration, the sponsor, the medical ethics committee of our hospital, the center ethics, and the office of drug clinical trial institution within 24 hours. When and by what means (e.g. telephone, fax or written) to whom SAE was reported should be recorded in the original data.
5. The original medical ethics committee reports the paper version, including the receipt page (with PI signature), SAE form and processing process in triplicate, and then reports the electronic version of PPT, which is then sent to wangxing5447@126.com
6. To study the doctor according to the implementation of treatment, if necessary, start to prevent and deal with medical subjects and emergency plans.
7. At the same time, the research doctor should make a record of SAE, including at least the description of adverse events, occurrence time, termination time, degree and frequency of seizures, and the treatment given.
8. The medical ethics committee will hold a meeting to organize experts to report and discuss the SAE and the treatment process in our hospital, and require the follow-up of SAE.

Sample size assessment

The purpose of this study was to verify whether the new strategy is not inferior to traditional method in uniport VATS upper lobe lobectomy. In terms of the incidence of pneumothorax (primary), based on previous observational studies, the probability of postoperative pneumothorax in new method and traditional method was about 10% and 6%. Considering 25% of non-inferiority margin, efficacy analysis estimated that 75 patients in each group were required to achieve power of 0.99 (via version 15.0; NCSs, Kaysville, UT, USA) with unilateral α of 0.025. Considering some out of groups due to clinical factors or other criteria (e.g., changing surgical methods according to pathological results during operation, combined with other lobectomy, etc.), a total of 75 subjects in each group were required, and 400 is the anticipating case number.

Plan for missing data The investigators made a plan for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results.

First, sufficient case is planned for the missing data generated from changes in surgery, as combined lobectomy or sublobectomies. Second, all the surgeons in our department will be informed of this study, and the changes in surgical method should be avoided to their best effort.

Statistical analysis plan

Statistical analysis will be performed to these select two groups in terms of clinical parameters, including the incidence of pneumothorax, reintubation rate, pain score and other parameters, respectively using t test, chi square test, rank sum test and other means. SPSS 20 will be validated to compare the primary and secondary observation end points between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uniport VATS for left / right upper lobectomy in Shanghai Pulmonary Hospital

Exclusion Criteria:

* preoperative presence of any unstable systemic disease, such as active infection, uncontrolled hypertension, or unstable angina pectoris;
* previous ipsilateral thoracic surgery;
* preoperative X-ray findings of pneumonia or atelectasis;
* bleeding tendency;
* anticoagulant use;
* pregnancy or breastfeeding;
* converted to open chest;
* the patient underwent pneumonectomy or segmental resection or wedge resection;
* severe adhesion occurred during the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
pneumothorax incidence | 24-30 hours after surgery
  The incidence of pneumothorax on day 1 after operation

SECONDARY OUTCOMES:
pain scores | 1day, 3days and 30 days after surgery
  pain scores collected after surgery
Extubation time | within 30 days after surgery
  Extubation time after operation
Total volume | 1 day after surgery
  Total volume of pleural effusion on the first day after operation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Gui, MD, Study Chair — Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mun M, Nakao M, Matsuura Y, Ichinose J, Nakagawa K, Okumura S. Video-assisted thoracoscopic surgery lobectomy for non-small cell lung cancer. Gen Thorac Cardiovasc Surg. 2018 Nov;66(11):626-631. doi: 10.1007/s11748-018-0979-x. Epub 2018 Jul 30. PMID 30062622
- [Result] Bulgarelli Maqueda L, Garcia-Perez A, Minasyan A, Gonzalez-Rivas D. Uniportal VATS for non-small cell lung cancer. Gen Thorac Cardiovasc Surg. 2020 Jul;68(7):707-715. doi: 10.1007/s11748-019-01221-4. Epub 2019 Oct 15. PMID 31617147
- [Result] Zhang JT, Dong S, Chu XP, Lin SM, Yu RY, Jiang BY, Liao RQ, Nie Q, Yan HH, Yang XN, Wu YL, Zhong WZ. Randomized Trial of an Improved Drainage Strategy Versus Routine Chest Tube After Lung Wedge Resection. Ann Thorac Surg. 2020 Apr;109(4):1040-1046. doi: 10.1016/j.athoracsur.2019.11.029. Epub 2020 Jan 8. PMID 31926158
- [Result] Liu CY, Hsu PK, Leong KI, Ting CK, Tsou MY. Is tubeless uniportal video-assisted thoracic surgery for pulmonary wedge resection a safe procedure? Eur J Cardiothorac Surg. 2020 Aug 1;58(Suppl_1):i70-i76. doi: 10.1093/ejcts/ezaa061. PMID 32182334